CLINICAL TRIAL: NCT04656678
Title: A Study to Evaluate the Safety and Efficacy of Focal US Guided Cryo-ablation Using DynaCAD / UroNAV Preplanning / Guidance of Locally Confined Low to Intermediate Risk Prostate Cancer
Brief Title: Focal US-guided Cryo-ablation Using DynaCAD / UroNAV Preplanning / Guidance of Intermediate Risk Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Ardeshir Rastinehad, Associate Professor of Urology and Radiology, Vice Chair of Urology at Lenox Hill Hospital, System Director for Prostate Cancer, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-0562
Record Dates: First submitted 2020-12-04; First posted 2020-12-07 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer; Prostate Disease
Keywords: Prostate MRI; Cryoablation; Focal Therapy; Focal Prostate Cancer Therapy; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- DynaCAD / UroNAV (Experimental): This is a single arm study to evaluate feasibility of UroNAV Ablation system aided cryo-ablation treatment of low and intermediate risk, organ-confined prostate cancer. UroNav is a stereotaxic accessory for image-guided interventional and diagnostic procedures of the prostate gland. It provides 2D and 3D visualization of Ultrasound (US) images and the ability to fuse and register these images with those from other imaging modalities such as Magnetic Resonance (MR), Computed Tomography, etc. It also provides the ability to display a simulated image of a tracked insertion tool on a computer monitor screen that shows images of the target organ and the current and the projected future path of the interventional instrument. DynaCAD 5.0 is an image analysis and planning system that will provide off station, pre planning and review of interventional study data. It interfaces with the Uronav 4.0 fusion guidance system.
  Interventions: Device: Cryo-ablation Using DynaCAD / UroNAV preplanning / guidance

INTERVENTIONS:
Device: Cryo-ablation Using DynaCAD / UroNAV preplanning / guidance — Focal ultrasound guided cryoablation using uroNav system Version 4.0 and Dyna CAD software version 5.0.

SUMMARY:
The purpose of this research study is to determine the safety and feasibility of using the UroNav software and DynaCAD software for planning and treating prostate cancer as an add on to the already approved workflow of using ultrasound only during the cryoablation of the prostate. The software application may aid doctors in locating a prior biopsy proven cancer location from the UroNav biopsy that patients previously had and then use that information to guide the treatment.

DETAILED DESCRIPTION:
This is a single-center, prospective, single arm study to evaluate feasibility of UroNAV Ablation system aided cryo-ablation treatment of low and intermediate risk, organ-confined prostate cancer. All subjects will be treated and then followed up clinically for up to 24 months to evaluate any procedure or device related adverse events as well as to assess efficacy endpoints of the study. Additional data related to quality of life of treated subjects will also be collected

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have documented histological or cytological evidence of tumor(s) of the prostate.
2. Patients must be ≥ 45 years of age.
3. Patients must be able to read, understand and sign an informed consent.
4. Organ confined clinical T1C or clinical T2a prostate cancer that is visualized on MR imaging.
5. Prostate cancer is diagnosed by MR image guided biopsies.
6. Gleason Score ≤ 7; and 2 or less positive lesions on prior MR US fusion guided prostate biopsy.
7. A non MRI visible cancer detected via systematic standard biopsy will not be considered an exclusion condition provided the non-MRI visible cancer is singularly located in the contralateral hemisphere of the prostate; is Gleason 6 cancer; and comprises no more than 6mm linear extent of cancer in a single core on standard biopsy.
8. If any standard biopsy cores are positive on the same hemisphere of the prostate gland, they must be confirmed as likely to form a contiguous lesion with the target lesion detected on MRI and therefore be from the same location in the prostate as MR lesion was biopsied and proven to be cancerous. (e.g., Left/Right, Base, Mid Gland, Apex).
9. Prior mpMRI results dated within 120 days prior to ablation.
10. No metastatic disease as per NCCN guidelines (www.nccn.org) - Bone scan indicated to r/o metastatic disease if clinical T1 and PSA > 20 or T2 and PSA > 10
11. PSA < 15 ng/ml or PSA density < 0.15 ng/ml2 in patients with a PSA > 15 ng/ml.

Exclusion Criteria:

1. ASA status > 3
2. Very Low Risk Prostate Cancer based on Epstein's Criteria having a tumor <0.2 cc (AUA Guidelines 2017 pg. 9)

   GG1, PSA < 10 ng/ml, no more than two positive cores and no core > 50% involvement.
3. Contraindications to MRI

   3.1 Claustrophobia

   3.2 Implanted ferromagnetic materials or foreign objects

   3.3 Known intolerance to the MRI or US contrast agents.

   3.4 Severely abnormal coagulation (INR>1.5)
4. Patients with unstable cardiac status including:

   4.1 Unstable angina pectoris on medication

   4.2 Patients with documented myocardial infarction within 40 days prior to enrolment

   4.3 Congestive heart failure NYHA class IV

   4.4 Patients with unstable arrhythmia status, already on anti-arrhythmic drugs
5. Severe hypertension (diastolic BP > 100 on medication)
6. Severe cerebrovascular disease (multiple CVA or CVA within 6 months)
7. History of orchiectomy, PCa-specific chemotherapy, brachytherapy, cryotherapy, Photodynamic therapy or radical prostatectomy for treatment of prostate cancer; any prior radiation therapy to the pelvis for prostate cancer or any other malignancy.
8. Patient under medications that can affect PSA for the last 3 months prior to UroNAV Ablation system aided cryo-ablation treatment (Androgen Deprivation Treatment)
9. Patients with lesions of Gleason 7 or greater outside the planned treatment area.
10. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (approximately 3 hrs.)
11. Any rectal pathology, anomaly or previous treatment, which could change acoustic properties of rectal wall or prevent safe US probe insertion (e.g., fistula, stenosis, fibrosis, inflammatory bowel disease, etc).
12. Any spinal pathology which can prevent safe administration of epidural/spinal anesthesia
13. Evidence for lymph node involvement of cancer
14. Bladder cancer
15. Urethral stricture/bladder neck contracture
16. Patients with incontinence demonstrated by use of more than 1 pad/day. .
17. Active UTI
18. Prostatitis NIH categories I, II and III.
19. Compromised renal function
20. Interest in future fertility
21. Current participation in another clinical investigation of a medical device or a drug or has participated in such a study within 30 days prior to study enrollment.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of safety of the DynaCAD /UroNAV ablation planning and guidance system aided cryo-ablation in the treatment of low-intermediate risk, localized (organ confined) prostate cancer tumors. | 24 months
  Incidence and severity of device/treatment related complications from treatment day visit through 24 month follow up.

SECONDARY OUTCOMES:
Assessment of tumor control achieved by treatment. | 24 months
  Primary effectiveness analyses will be based on the 12-month biopsy results. Post-treatment PSA, non-perfused volume (NPV) by multi-parametric MRI, and EPIC - 26 (The Expanded Prostate Cancer Index Composite) questionnaire results through Month 24 visit will be summarized as secondary measures of effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Ardeshir Rastinehad, DO, Principal Investigator — Northwell Health
Locations (3):
- United States (3):
  - The Smith Institute for Urology, Lake Success, New York
  - The Smith Institute for Urology at Lenox Hill, New York, New York
  - Manhattan Eye, Ear, and Throat Hospital (MEETH), New York, New York

REFERENCES:
- [Derived] Jue JS, Coons S, Hautvast G, Thompson SF, Geraats J, Richstone L, Schwartz MJ, Rastinehad AR. Novel Automated Three-Dimensional Surgical Planning Tool and Magnetic Resonance Imaging/Ultrasound Fusion Technology to Perform Nanoparticle Ablation and Cryoablation of the Prostate for Focal Therapy. J Endourol. 2022 Mar;36(3):369-372. doi: 10.1089/end.2021.0266. Epub 2021 Sep 13. PMID 34409850